CLINICAL TRIAL: NCT04011046
Title: Register of Patients Benefiting From a Coronary Bifurcation Angioplasty at the University Hospital of Nîmes and Montpellier in 2017
Acronym: Register
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2017
Record Dates: First submitted 2019-07-01; First posted 2019-07-08 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Stent Thrombosis
MeSH Terms: interventions — Stents

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Stent

SUMMARY:
Cardiovascular diseases are the second leading cause of death in France and the world's leading cause.Coronary bifurcations are conducive to the development of atheromatous lesions due to flow turbulence generating a pro-atherogenic effect. They represent about 15% of coronary lesions and 30% of lesions in pluri truncular patients.Coronary bifurcation angioplasty is a complex angioplasty with a high risk of complications.Numerous studies have compared different angioplasty techniques with 2 stents in bifurcation lesions. However, two studies of The Nordic-Baltic Bifurcation Study did not show at 6 months or 5 years of age any significant difference in major cardiovascular events (death, heart attack, stent thrombosis, emergency revascularization of the target vessel) in patients with a one-stent strategy compared to the systematic use of two stents. There are also several post-expansion techniques and the one that appears to be the most commonly used today (known as the "KISSING-BALLOON") consists of inflating two balloons at the same time, one in the main branch and the other in the daughter branch in order to open the meshes of the stent towards the daughter branch. Studies on a test bench to evaluate the deformation of a stent in different coronary anatomies according to the material and technique used have nevertheless revealed several limitations to this technique, in particular an elliptical deformation of the stent linked to the inflation of 2 simultaneous balloons.

From this work, a new technique known as "POT SIDE POT" was born, consisting in post dilating the proximal part of the stent of the main branch in order to place it as closely as possible against the wall, then open the stent meshes towards the lateral branch by balloon dilation followed by a new post dilation of the proximal part of the mother branch stent to avoid the use of 2 simultaneous balloons and thus reduce stent deformation by maintaining a circular geometry while allowing proper stent attachment.

However, to date, there are no clinical studies comparing the POT SIDE POT technique with that of KISSING-BALLOON in coronary bifurcation angioplasty.

This is why we would like to compare these two post-dilation techniques by a retrospective study on the occurrence of major cardiovascular events and stent thrombosis in patients who received a coronary bifurcation angioplasty in 2017 at the University Hospital of Nîmes.

DETAILED DESCRIPTION:
Cardiovascular diseases are the second leading cause of death in France and the world's leading cause.Coronary bifurcations are conducive to the development of atheromatous lesions due to flow turbulence generating a pro-atherogenic effect. They represent about 15% of coronary lesions and 30% of lesions in pluri truncular patients.Coronary bifurcation angioplasty is a complex angioplasty with a high risk of complications.Numerous studies have compared different angioplasty techniques with 2 stents in bifurcation lesions. However, two studies of The Nordic-Baltic Bifurcation Study did not show at 6 months or 5 years of age any significant difference in major cardiovascular events (death, heart attack, stent thrombosis, emergency revascularization of the target vessel) in patients with a one-stent strategy compared to the systematic use of two stents. There are also several post-expansion techniques and the one that appears to be the most commonly used today (known as the "KISSING-BALLOON") consists of inflating two balloons at the same time, one in the main branch and the other in the daughter branch in order to open the meshes of the stent towards the daughter branch. Studies on a test bench to evaluate the deformation of a stent in different coronary anatomies according to the material and technique used have nevertheless revealed several limitations to this technique, in particular an elliptical deformation of the stent linked to the inflation of 2 simultaneous balloons.

From this work, a new technique known as "POT SIDE POT" was born, consisting in post dilating the proximal part of the stent of the main branch in order to place it as closely as possible against the wall, then open the stent meshes towards the lateral branch by balloon dilation followed by a new post dilation of the proximal part of the mother branch stent to avoid the use of 2 simultaneous balloons and thus reduce stent deformation by maintaining a circular geometry while allowing proper stent attachment.

However, to date, there are no clinical studies comparing the POT SIDE POT technique with that of KISSING-BALLOON in coronary bifurcation angioplasty.

This is why we would like to compare these two post-dilation techniques by a retrospective study on the occurrence of major cardiovascular events and stent thrombosis in patients who received a coronary bifurcation angioplasty in 2017 at the University Hospital of Nîmes.

ELIGIBILITY:
Inclusion Criteria:

* All angioplasties of bifurcation lesion to a de novo stent defined by :
* MEDINA classification 1,1,1,1 or 0,1,1,1 or 1,0,1
* Diameter of the mother and daughter branch > 2.5mm
* No history of angioplasty of this bifurcation (de novo lesion)
* Accessible for coronary angioplasty treatment
* Patients admitted to the University Hospital of Nîmes from January 1 to December 31, 2017

Exclusion Criteria:

* Minor patient
* Bifurcation lesion not meeting the above criteria
* Cardiorespiratory arrest
* Injury on bypass surgery
* Intrastent restenosis
* 2-stent angioplasty technique

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * All angioplasties of bifurcation lesion to a de novo stent defined by :
  * MEDINA classification 1,1,1,1 or 0,1,1,1 or 1,0,1
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of a composite criterion associating major ischemic events (Major adverse Cardiac Events: death from any cause, myocardial infarction, need for revascularization) and the occurrence of stent thrombosis during hospitalization. | within one year
  Occurrence of a composite criterion associating major ischemic events (Major adverse Cardiac Events: death from any cause, myocardial infarction, need for revascularization) and the occurrence of stent thrombosis during hospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nîmes, Nîmes, France